CLINICAL TRIAL: NCT03739593
Title: A Multicenter, Open-label, Safety and Proof-of-concept Study to Assess Safety, Tolerability and Efficacy of AR-1105 in Subjects With Macular Edema Due to Retinal Vein Occlusion (RVO)
Brief Title: Study Assessing AR-1105 in Subjects With Macular Edema Due to Retinal Vein Occlusion (RVO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR-1105-CS201
Record Dates: First submitted 2018-11-08; First posted 2018-11-14 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Macular Edema
Keywords: Macular Edema; Retinal Vein Occlusion; Dexamethasone Intravitreal Implant
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Single injection of either of 2 formulations of AR-1105 dexamethasone intravitreal implant (CF1 or CF2) administered in a single eye. An initial safety cohort of up-to 5 subjects may be enrolled onto CF1 prior to the randomized phase. During the randomized phase of the study, subjects will be assigned in a 1:1 ratio to either CF1 or CF2. Each subject will complete a 6-month primary evaluation period. Residual implant assessment will be performed by 3-field fundus photography at Day 7 and at Months 3, 4, 5, and 6, and if necessary at monthly visits thereafter until the subject requires retreatment, or until 1 month after the implant is no longer visible, or to Month 9, whichever comes first.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AR-1105-CF1 (Experimental): Single dose of AR-1105-CF1 (dexamethasone, targeted dose of 340 mcg) administered as an intravitreal implant into a single eye of up to 20 subjects who will be followed for 6 months
  Interventions: Drug: AR-1105-CF1
- AR-1105-CF2 (Experimental): Single dose of AR-1105-CF2 (dexamethasone, targeted dose of 340 mcg) administered as an intravitreal implant into a single eye of up to 20 subjects who will be followed for 6 months
  Interventions: Drug: AR-1105-CF2

INTERVENTIONS:
Drug: AR-1105-CF1 — AR-1105 clinical formulation 1 (AR-1105-CF1)
  Other Names: AR-1105-CF1 (dexamethasone intravitreal implant)
  Arms: AR-1105-CF1
Drug: AR-1105-CF2 — AR-1105 clinical formulation 2 (AR-1105-CF2)
  Other Names: AR-1105-CF2 (dexamethasone intravitreal implant)
  Arms: AR-1105-CF2

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of AR-1105 (dexamethasone implant) for the treatment of macular edema (ME) due to retinal vein occlusion (RVO). A more durable intravitreal implant containing a low dose of dexamethasone may result in less frequent retreatments, and potentially lower the incidence of steroid-related side effects without compromising efficacy.

DETAILED DESCRIPTION:
AR-1105 is a dexamethasone containing implant drug delivery system that is injected into the back of the eye. It is designed to dissolve slowly over time, continuously releasing a consistent low dose of steroid to treat the symptoms of RVO and associated inflammation with a goal of halting further visual disturbance and damage, and also possibly restoring some vision as symptoms are controlled. In this study, 2 different formulations are being tested to find the optimum combination of efficacy, safety and durability that will offer patients a potential treatment option that is as safe and effective as the treatments currently available, but which requires less frequent injections and potentially has a lower risk for certain side-effects.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Vision loss due to clinically detectable macular edema (ME) associated with either central retinal vein occlusion (CRVO) or branch retinal vein occlusion (BRVO). Subjects may be treatment-naïve, or if previously-treated with a steroid, must have demonstrated response to treatment
3. Duration of macular edema (ME) ≥9 months in subjects with CRVO and ≥12 months in subjects with BRVO. If both eyes are eligible, the study eye will be the eye with worse VA
4. Best-corrected visual acuity (BCVA) as measured by the early treatment of diabetic retinopathy study (ETDRS) methodology of between 25 and 70 letters, in the study eye and better than 35 letters, in the non-study eye
5. Retinal thickness in the central subfield of >290 µm (females) and >305 μm (males) if using a Cirrus (Zeiss) instrument, or if a Spectralis (Heidelberg) instrument is used, thickness should be >305 μm (females) or >320 μm (males) in the study eye
6. Be able to understand and willing to provide written informed consent.
7. Be willing and able to adhere to the instructions set forth in the study protocol

Exclusion Criteria:

Ophthalmic:

1. Presence of a clinically significant epiretinal membrane, active retinal or optic disc neovascularization, active or history of choroidal neovascularization, presence of rubeosis iridis
2. History or presence of herpetic infection, toxoplasmosis, chorioretinopathy.
3. Subjects with moderate non-proliferative diabetic retinopathy or worse in either eye are excluded from participation
4. Any active infection
5. Aphakia, significant posterior capsule tear or iris trauma in the study eye
6. Anterior-chamber intraocular lens
7. Clinically significant media opacity
8. History of glaucoma or visual field loss
9. Ocular hypertension in the study eye at qualification, (with or without treatment)
10. History of corticosteroid-induced IOP increase in either eye
11. Ocular condition in the study eye that, in the opinion of the investigator, would prevent a 15-letter improvement in visual acuity
12. Received an intraocular steroid injection or implant within 6 months or any anti-VEGF treatment within 2 months prior to screening. Prior treatment with RETISERT® or ILUVIEN® or pan-retinal photocoagulation (PRP) is exclusionary
13. Intraocular surgery (including laser refractive or eyelid surgery) within 3 months prior to Visit 1 or anticipated need for ocular surgery or ophthalmic laser treatment during the study treatment period
14. Currently using topical corticosteroids in the vicinity of the eyes within the 1 month prior to Visit 1
15. Periocular depot of steroids placed within 6 months prior to qualification
16. Ocular medications that are specifically disallowed in this protocol for any condition during the study or within the specified timeframe prior to Visit 2
17. Have progressive optic nerve disease or retinal disease other than retinopathy due to RVO that affects BCVA

    Systemic:
18. Currently using or anticipating the use of systemic corticosteroids during the study (with the exception of inhaled, intranasal or topical corticosteroids)
19. Any clinically significant or uncontrolled serious or severe medical or psychiatric condition
20. Participation in any other interventional clinical study within 30 days prior to Visit 1
21. History of hypersensitivity or poor tolerance to any components of the preparations to be used in this study such as dexamethasone or biodegradable polymer (PLGA) excipients or fluorescein
22. Systemic condition that may confound the study outcome per the investigator's opinion
23. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rowan, Study Director — Aerie Pharmaceuticals, Inc.
Locations (11):
- United States (11):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina Vitreous Associates, Beverly Hills, California
  - Byers Eye Institute at Stanford, Palo Alto, California
  - Florida Eye Clinic, Altamonte Springs, Florida
  - Center for Retina & Macular Disease, Lakeland, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Mid-Atlantic Retina, Cherry Hill, New Jersey
  - Cleveland Clinic- Cole Eye Institute, Cleveland, Ohio
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singer MA, Boyer DS, Williams S, McKee H, Kerr K, Pegoraro T, Trevino L, Kopczynski CC, Hollander DA. PHASE 2 RANDOMIZED STUDY (ORION-1) OF A NOVEL, BIODEGRADABLE DEXAMETHASONE IMPLANT (AR-1105) FOR THE TREATMENT OF MACULAR EDEMA DUE TO CENTRAL OR BRANCH RETINAL VEIN OCCLUSION. Retina. 2023 Jan 1;43(1):25-33. doi: 10.1097/IAE.0000000000003632. Epub 2022 Oct 14. PMID 36542081

RESULTS

PARTICIPANT FLOW:
Groups:
- Initial Phase: AR-1105-CF1; Randomization Phase: AR-1105-CF1: Single dose of AR- 1105-clinical formulation 1 (CF1) dexamethasone 340 mcg administered as an intravitreal implant into a single eye
- Randomization Phase: AR-1105-CF2: Single dose of AR- 1105-clinical formulation 2 (CF2) dexamethasone 340 mcg administered as an intravitreal implant into a single eye
Period: Overall Study
Arm/Group | Initial Phase: AR-1105-CF1 | Randomization Phase: AR-1105-CF1 | Randomization Phase: AR-1105-CF2
Started | 5 | 22 | 22
Completed | 2 | 16 | 14
Not Completed | 3 | 6 | 8

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- AR-1105-CF1 Initial Phase; AR-1105-CF1 Randomization Phase: Single dose of AR-1105-CF1 (dexamethasone 340 mcg) administered as an intravitreal implant into a single eye
- AR-1105-CF2 Randomization Phase: Single dose of AR-1105-CF2 (dexamethasone, 340 mcg) administered as an intravitreal implant into a single eye
- Total: Total of all reporting groups
Arm/Group | AR-1105-CF1 Initial Phase | AR-1105-CF1 Randomization Phase | AR-1105-CF2 Randomization Phase | Total
Number analyzed (Participants) | 5 | 22 | 22 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 10 | 6 | 18
  >=65 years | 3 | 12 | 16 | 31
Age, Continuous [Median (Full Range); unit: Years] | 67 [57 to 87] | 66 [27 to 88] | 72 [47 to 88] | 68 [27 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 9 | 13 | 22
  Male | 5 | 13 | 9 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : American Indian or Alaska Native | 0 | 1 | 0 | 1
  Race : Asian | 0 | 0 | 2 | 2
  Race : Black or African American | 0 | 2 | 1 | 3
  Race : Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race : White | 5 | 19 | 19 | 43
  Race : Other | 0 | 0 | 0 | 0
  Race : Multiple Race | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 22 | 22 | 49

OUTCOME MEASURES:

1. Primary Outcome: Safety Tolerability: Number of Ocular and Non-ocular TEAEs
Description: Treatment-emergent adverse events summarized at the subject level by system organ class and preferred term are available in the Adverse Events module. Data reported in the table below corresponds to the total number of participants with ocular and non-ocular treatment-emergent adverse events (TEAEs).
Time Frame: Up to 6 months treatment duration
Population: All safety evaluations were conducted on subjects in the safety population. The safety population included all subjects who received study medication. This population was used to summarize safety variables. Subjects were analyzed as-treated
Measure: Number; unit: participants
Groups:
- Initial Phase: AR-1105-CF1; Randomization Phase: AR-1105-CF1: Single dose of AR-1105-clinical formulation 1 (CF1) dexamethasone 340 mcg administered as an intravitreal implant into a single eye
- Randomization Phase: AR-1105-CF2: Single dose of AR-1105-clinical formulation 2 (CF2) dexamethasone 340 mcg administered as an intravitreal implant into a single eye
Arm/Group | Initial Phase: AR-1105-CF1 | Randomization Phase: AR-1105-CF1 | Randomization Phase: AR-1105-CF2
Number analyzed (Participants) | 5 | 22 | 22
participants | 5 | 22 | 22

ADVERSE EVENTS:
Time Frame: Adverse events were documented from the time the subject signed the informed consent until Month 6 + 30 days, or up to Month 9 + 30 days in subjects with visible residual implant observed at Month 6 or beyond.
Groups:
- Randomization Phase: AR-1105-CF2: Single dose of AR- 1105-clinical formulation 1 (CF2) dexamethasone 340 mcg administered as an intravitreal implant into a single eye
Arm/Group | Initial Phase: AR-1105-CF1 | Randomization Phase: AR-1105-CF1 | Randomization Phase: AR-1105-CF2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/22 | 4/22
Other Adverse Events (participants affected / at risk) | 5/5 | 9/22 | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Phase: AR-1105-CF1 (N=5) | Randomization Phase: AR-1105-CF1 (N=22) | Randomization Phase: AR-1105-CF2 (N=22)
Visual Acuity Reduced (Eye disorders) | 1 | 1 | 2
Iris Neovascularization (Eye disorders) | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Visual Impairment (Eye disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Phase: AR-1105-CF1 (N=5) | Randomization Phase: AR-1105-CF1 (N=22) | Randomization Phase: AR-1105-CF2 (N=22)
Visual Acuity Reduced (Eye disorders) | 1 | 2 | 3
Macular Edema (Eye disorders) | 2 | 4 | 2
Conjunctival Haemorrhage (Eye disorders) | 2 | 2 | 1
Ocular Hypertension (Eye disorders) | 0 | 0 | 3
Vitreous Haemorrhage (Eye disorders) | 0 | 0 | 3
Vitreous Floaters (Eye disorders) | 0 | 0 | 2
Intraocular Pressure Increased (Investigations) | 1 | 1 | 3
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0
Device Malfunction (Product Issues) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT03739593/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT03739593/SAP_001.pdf